CLINICAL TRIAL: NCT07361614
Title: Pilot Testing of a Colorectal Cancer Education Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25-01040; K01CA255411 (NIH)
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer Screening
Keywords: CRC; Colorectal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults due for CRC screening who speak English or a Chinese language (Cantonese/Mandarin) (Experimental): Participants will receive one CRC educational session, which will take around 1-1.5 hours.
  Interventions: Behavioral: Educational Program

INTERVENTIONS:
Behavioral: Educational Program — Culturally and linguistically tailored program consisting of community health worker (CHW)-led education sessions followed by patient navigation (PN) services.

SUMMARY:
The primary objective of this study is to assess the feasibility, acceptability, and preliminary efficacy of a culturally and linguistically targeted, colorectal cancer (CRC) education program to improve CRC screening completion.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-75 years
2. Not guideline concordant (no stool testing for CRC within past 1 year)
3. No colonoscopy in past 10 years; no sigmoidoscopy or CT colonography in past 5 years)
4. Understands English or Chinese languages.
5. Willing and able to consent to participate

Exclusion Criteria:

1) history of CRC or colectomy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
CRC screening completion (yes/no) | Month 6

SECONDARY OUTCOMES:
Change in Brief Illness Perception Questionnaire (IPQ-B) score | Baseline, Month 6
  The IPQ-B is a 9-item questionnaire (validated in the Chinese population) that assesses CRC beliefs according to CRC beliefs according to SRM constructs (SRM) constructs. Each item is rated on a scale from 0 (strong disagree) to 10 (strongly agree). Total scores range from 0-90, with higher scores indicating a greater threat and worse perception of illness.
Change in Medicines Questionnaire (BMQ) score | Baseline, Month 6
  The BMQ, validated in the Chinese population, adapted to assess concerns/necessity of CRC screening is a 5 items questionnaire. Items are assessed on a scale from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 5-25, with higher scores indicating positive beliefs about CRC screening.
Change in number of barriers to care | Baseline, Month 6
  Participants re asked to select all that apply to barriers in care: Cost, Transportation, Lack of time, Fear of results, Embarrassment, Lack of trust in doctors, Language barriers, Other. Each item selected is counted, a decrease in the number of items selected indicates reduced barriers to care.
Change in trust in health/community health workers | Baseline, Month 6
  Group-based medical mistrust scale consists of 2 statements of mistrust and 2 statements of trust. Each statement can be answered with 1) Strongly Disagree, 2) Disagree, 3) Neither Agree nor Disagree, 4) Agree, 5) Strongly Agree.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Vang, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to Suzanne.vang@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Suzanne.vang@nyulangone.org To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.